CLINICAL TRIAL: NCT01980212
Title: Serum Thioredoxin Reductase Activity Research in First-line Chemotherapy Advanced Non-small Cell Lung Cancer
Brief Title: Tumor Relapsed Study of Serum Trxr Activity in Advanced Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, chief, Hunan Province Tumor Hospital
Other Study IDs: TRSTILC
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Advanced Non-small Cell Lung Cancer; First Line Treatment; Thioredoxin Reductase Activity; Carcinoembryonic Antigen; Progression
Keywords: non-small cell lung cancer; thioredoxin reductase
MeSH Terms: conditions — Disease Progression; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3-4 ml whole blood was obtained and then centrifuged and stored at -20 ℃
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- first line advanced non-small cell lung cancer: patients newly diagnosed advanced non-small cell lung cancer, and received platinum based chemotherapy in Hunan Province Tumor Hospital

SUMMARY:
In pre-clinical study we found that the thioredoxin reductase activity of serum harbours huge difference between cancer patients and non-cancer patients, the enzyme activity elevated remarkably among cancer patients, and after any kind of treatment serum thioredoxin reductase activity declined remarkably, so we hypothesis that serum thioredoxin reductase activity could be a warning marker for early progression of first-line treatment for advanced non-small cell lung cancer

DETAILED DESCRIPTION:
This is a cooperative research project involving patients in Medical Oncology Department of Affiliated Cancer Hospital of Xiangya School of Medicine Central South University, and the State Key Laboratory for Natural Medicine and Biomimetic Drugs Perking University. The primary objective is to measure the thioredoxin reductase activity using blood in subjects received platinum based chemotherapy, to study the warning progression ability of thioredoxin reductase in blood. The secondary objective is to compare the warning progression activity of blood thioredoxin reductase reductase activity with carcinoembryonic antigen in subjects received platinum based first-line chemotherapy. Blood will be collected before chemotherapy, after every 2 cycles of chemotherapy, every 3 months after all first-line chemotherapy till 2 years, then every 6 months till 3 years, or collect blood till tumor progression, evaluation CT results every time collecting blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven non-small cell lung cancer, stage Ⅳ patients or unsuitable for local treatment of ⅢB stage patients
* Malignant tumor treatment naive including surgery（except for surgery for cervical cancer and cutaneous squamous cell carcinoma 5 years before, except for lung cancer patients who received surgery and adjuvant chemotherapy after 12 month then diagnosed with stage ⅢB or Ⅳ）
* Signed informed consent would like to provide blood for research

Exclusion Criteria:

* Patients received antitumor treatment before
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-small lung cancer and receiving platinum based first-line chemotherapy in Medical Oncology Department of Affiliated Cancer Hospital of Xiangya School of Medicine Central South University/Hunan Province Tumor Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
To measure the thioredoxin reductase activity in blood | may 2013 - may 2014 (1 year)
  3-4 ml whole blood was obtained and then centrifuged and stored at -20 ℃, thioredoxin reductase activity was measured within 30 days using 5，5'-Dithio bis-（2-nitrobenzoic acid）(DTNB) method.

SECONDARY OUTCOMES:
To measure the carcinoembryonic antigen (CEA) level in blood | may 2013- may 2014 (1 year)
  Measure the CEA level every time compared with thioredoxin reductase activity

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Study Chair — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China